CLINICAL TRIAL: NCT00533455
Title: A 4 Week, Parallel-Design, Double-Blind, Placebo-Controlled Trial of Gabapentin in the Treatment of Neuroleptic-Induced Tremor: Clinical and Instrumental Ratings of Outcome.
Brief Title: Gabapentin for the Treatment of Neuroleptic-Induced Tremor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to recruit due to polypharmacy
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3232-A
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Neuroleptic-Induced Tremor
Keywords: Antipsychotics, tremor
MeSH Terms: conditions — Tremor | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gabapentin

SUMMARY:
We will attempt to establish whether gabapentin as compared with placebo will reduce the severity of tremors caused by the use of antipsychotic medications. Baseline severity of tremor will be measured using both clinical ratings and ratings obtained with an instrument designed to measure tremor, giving more objective evidence of tremor frequency and severity.

DETAILED DESCRIPTION:
We propose to enroll 40 veterans with antipsychotic induced tremor in this RCT of gabapentin. Baseline measurements will be obtained with the tremor section of the UPDRS, the Simpson-Angus Scale, the ESRS, AIMS, and the Barnes Akathisia SScale. The Tremorometer, an instrument designed to quantatatively measure frequency, amplitude, and tremor power will be used for baseline and subsequent assessments. Demographic data will be collected. Diagnoses will be established with the SCID. Appropriate lab studies with an EKG will be done at baseline and at study end. Patients will be randomized to gabapentin or placebo and assessed on a blinded basis. Effectiveness of the blind will be assessed at study end. Gabapentin will be started at 300 mg/day and tapered up to a maximum of 1800 mg/day. The SF36 will be used to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 18 and older with an observable tremor judged to be caused by exposure to antipsychotics

Exclusion Criteria:

* Concomitant use of other anticonvulsants, L-Dopa, cocaine, amphetamines, or other tremorogenic agents excepting SSRIs, TCAs.
* Current suicidality, severe psychosis, inability to sign informed consent or to cooperate with study procedures.
* Current use of gabapentin or exposure to gabapentin in the past 2 years.
* Women who are pregnant, or not using adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Reduction of tremor on the UPDR and SAS
Reduction of instrumental measurements of percent tremor and tremor power.

SECONDARY OUTCOMES:
Reduction of rigidity, bradykinesia, dyskinesia
Improvement in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Dean, MD, Principal Investigator — Minneapols VA Medical Center; Adityanjee Adityanjee, MD, Study Director — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapols VA Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Onofrj M, Thomas A, Paci C, D'Andreamatteo G. Gabapentin in orthostatic tremor: results of a double-blind crossover with placebo in four patients. Neurology. 1998 Sep;51(3):880-2. doi: 10.1212/wnl.51.3.880. PMID 9748048